CLINICAL TRIAL: NCT07177508
Title: First Year Impact of Nirsevimab on Paediatric Respiratory Syncytial Virus Infection and Hospitalisations in the Australian Capital Territory: An Observational Study
Brief Title: First Year Impact of Nirsevimab on Paediatric Respiratory Syncytial Virus Infection and Hospitalisations in the Australian Capital Territory
Status: Completed | Type: Observational
Sponsor: Nicola Irwin (Other)
Responsible Party: Sponsor-Investigator, Nicola Irwin, Principal Investigator, The Canberra Hospital
Organization: The Canberra Hospital (Other)
Other Study IDs: 2024.LRE.00283
Record Dates: First submitted 2025-09-10; First posted 2025-09-17 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Respiratory Syncytial Viral (RSV) Infection; Respiratory Syncytial Virus Hospitalizations; Respiratory Syncytial Virus Prevention
Keywords: Epidemiological Methods; Infections
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- RSV cases: Children under 2 years of age with laboratory confirmed RSV infection

SUMMARY:
The goal of this observational study is to explore the impact of a new prevention medicine (nirsevimab) on the burden of Respiratory Syncytial Virus (RSV) disease in children under 2 years of age. The main question it aims to answer is:

How has the incidence of RSV, and Emergency Department presentations and hospital admissions for RSV-related disease changed since nirsevimab was introduced? Participants won't need to do anything extra for this research study, as only routinely collected data will be used for analysis.

DETAILED DESCRIPTION:
RSV infection is the leading cause for hospitalisation in young children. Treatment of RSV is primarily supportive, and includes supplemental oxygen therapy, ventilatory support, and fluid management. Prevention of paediatric RSV has been limited to monoclonal antibody (MAB) use for selected high-risk infants: palivizumab, a neutralising antibody against RSV, reduces RSV-related hospitalisation and illness severity in high-risk infants when administered monthly throughout the RSV season. Palivizumab was approved in Australia in 1999, however cost effectiveness has curtailed broad access. A novel long-acting monoclonal antibody, nirsevimab, was approved in Australia in November 2023. A single dose provides protection against RSV for the duration of an RSV season, and it is now recommended in preference to palivizumab. Nirsevimab is funded by individual jurisdictions. The Australian Capital Territory (ACT) commenced a nirsevimab program in April 2024, offered to infants born less than 37 weeks' gestation after 31st October 2023, all Aboriginal and Torres Strait Islander babies born after 31st October 2023, and infants with specific medical conditions.

This study aims to describe and compare the incidence of RSV infection, RSV-related ED presentations and hospital admissions, and severity of illness in children <2 years in the ACT, pre- and post- nirsevimab introduction. he pre-nirsevimab period will be defined as 1/4/2022 to 31/3/2024 and the post-nirsevimab period 1/4/2024 to 31/3/2025.

ELIGIBILITY:
Inclusion Criteria:

* child aged less than 2 years
* laboratory confirmed RSV

Exclusion Criteria:

* n/a

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study is set in the Australian Capital Territory, a small Australian jurisdiction with a single acute paediatric service provider.
Sampling Method: Non-Probability Sample
Enrollment: 2355 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
RSV hospitalisation | Over a period of 3 years
  RSV-related hospital admissions will be determined by reviewing hospital admissions occurring within one month of a positive RSV test. The discharge summary will be reviewed for a diagnosis or other clinical information consistent with RSV-related illness (bronchiolitis, respiratory tract infection, viral illness), and cross-checked with the ICD-10-AM coding for the episode.
RSV cases | Over a period of 3 years
  RSV cases will be determined by laboratory notifications of positive RSV infection on PCR test to ACT Health, the body responsible for receiving notifiable disease notifications.
Emergency Department presentations | Over a period of 3 years
  RSV-related ED presentations will be determined by reviewing ED presentations occurring within one month of a positive RSV test. Documentation from the presentation will be reviewed for a discharge diagnosis or impression consistent with RSV-related illness (bronchiolitis, respiratory tract infection, viral illness). If no discharge letter or doctors' documentation is available, the triage note will be reviewed for a presenting complaint consistent with RSV-related illness (rhinorrhoea, nasal congestion, cough, respiratory distress, diffuse crackles and/or wheeze, fever, hypoxaemia, and associated feeding difficulties, vomiting, dehydration, or lethargy).

CONTACTS AND LOCATIONS:
Locations (1):
- The Canberra Hospital, Garran, Australian Capital Territory, Australia

IPD SHARING:
Plan to Share IPD: Yes
Deidentified IPD that underlie any published results may be shared upon reasonable request, and subject to ethics and governance processes
Supporting Information: Study Protocol
Time Frame: From 3 months after publication of results to 3 years.
Access Criteria: Researchers with a methodologically sound proposal, subject to ethics and governance processes. A data sharing agreement will be required.
URL: https://www.act.gov.au/open/act-data-sharing-policy